CLINICAL TRIAL: NCT06564480
Title: A Prospective, Randomized, Parallel Controlled, Non Inferiority Clinical Trial Evaluating the Effectiveness and Safety of the Walker Assisted Device (Fubon Robot) in Lower Limb Motor Function for Stroke Patients
Brief Title: A Study on the Effectiveness Evaluation in Stroke Patients Using Lower Limb Assistive Walking Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang Hospital (Other); Zhejiang Provincial Tongde Hospital (Other); Zhejiang University (Other); Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-205
Record Dates: First submitted 2024-08-14; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Stroke
Keywords: stroke; Lower Extremity; Walking
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): Patients received MI-R1 lower limb walking machine assisted training device based on their condition for the following training content:
  1. Center of gravity transfer training;
  2. Marking time and walking training;
  3. Transfer training; 15 minutes each time, once a day, at least 5 times a week.
  Interventions: Device: MI-R1 lower limb walking machine assisted training device
- control group (Active Comparator): Patients received walking rehabilitation training under the guidance of therapists based on their condition for the following training content:
  1. Center of gravity transfer training;
  2. Single leg weight-bearing training;
  3. Marking time training assisted by balance bar；
  4. Walking training assisted by balance bar; 15 minutes each time, once a day, at least 5 times a week.
  Interventions: Other: Walking rehabilitation training under the guidance of therapists

INTERVENTIONS:
Device: MI-R1 lower limb walking machine assisted training device — The training is conducted under partial weight support training conditions, performing passive movements on the lower limbs through motor drive, improving the joint activity of the patient's hip and knee joints, and achieving sitting, standing, and walking functions.
  Arms: treatment group
Other: Walking rehabilitation training under the guidance of therapists — Each patient undergoes training under the guidance of a rehabilitation therapist
  Arms: control group

SUMMARY:
The main purpose of this clinical trial is to evaluate the effectiveness and safety of the MI-R1 walking machine in lower limb motor function training for stroke patients.

The main question is to answer:

1. Are patients using MI-R1 lower limb walking machine training more effective than those using traditional rehabilitation training?
2. Is the MI-R1 lower limb walking machine safe?

Participants will:

1. The experimental group received MI-R1 lower limb walking machine assisted training, while the control group received traditional rehabilitation training.
2. Perform functional testing on the 0th, 14th, and 28th day of training.
3. Observe whether there is any discomfort or safety during the rehabilitation training process.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with stroke through CT or MRI, and only accompanied by hemiplegia on one side, with first-time onset or previous episodes without residual neurological dysfunction;
* Vital signs stable, neurological symptoms no longer aggravate after 48 hours, no severe cognitive impairment or aphasia, and cooperate with training;
* Modified Ashworth score for lower limb ≤ level 2, standing balance function level ≥1;
* Voluntarily participating in this trial, understanding and cooperating with the entire trial process, and signing a written informed consent form.

Exclusion Criteria:

* Bone, joint, muscle disease, or lower limb disabilities (such as severe osteoporosis, fractures, spinal instability, severely limited joint range of motion, severe limb muscle contractures, deformities, etc.) or diseases that affect balance and walking;
* Stroke caused by cerebellar brainstem injury and cortical injury;
* Patients with severe primary diseases such as cardiovascular, pulmonary, hepatic, renal, and hematopoietic systems, as well as critically ill and psychiatric patients;
* Other contraindications or complications that may affect walking training treatment;
* Patients with local skin damage or pressure ulcers in the lower limbs;
* Patients with peripheral nerve injury in the lower limbs;
* Inappropriate body shape for robots (height<150cm or>190cm, or weight>85 kg);
* Planned pregnancy or pregnant and lactating women;
* Participants in other clinical trials within the past 3 months;
* Severe cognitive impairment;
* Known refusal or inability to comply with protocol requirements for any reason (including planned clinical visits and examinations);
* The researchers believe that it should not participate in this clinical trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Fugl Meyer Lower Limb Balance Assessment Scale Score on the 28th day | through study completion, an average of one and a half year
  Lower limb function assessment

SECONDARY OUTCOMES:
Fugl Meyer Lower Limb Balance Assessment Scale Score on the 0th and 14th day | through study completion, an average of one and a half year
  Lower limb function assessment
Holden Walking Function Classification | through study completion, an average of one and a half year
  Pedestrian function assessment on the 0th，14th and 28th day
Modified Barthel Index | through study completion, an average of one and a half year
  Assessment of activities of daily living ability on the 0th，14th and 28th day

OTHER OUTCOMES:
Vital signs - temperature | through study completion, an average of one and a half year
  Measure the patient's body temperature on the 0th, 14th, and 28th days of training
Vital signs - heart rate | through study completion, an average of one and a half year
  Measure the patient's heart rate on the 0th, 14th, and 28th days of training
Vital signs - respiratory rate | through study completion, an average of one and a half year
  Measure the patient's respiratory rate on the 0th, 14th, and 28th days of training
Vital signs - blood pressure | through study completion, an average of one and a half year
  Measure the patient's blood pressure on the 0th, 14th, and 28th days of training
Vital signs - pulse | through study completion, an average of one and a half year
  Measure the patient's pulse on the 0th, 14th, and 28th days of training
Adverse events | through study completion, an average of one and a half year
  Number of participants with treatment-related adverse events as assessed by "Criteria for determining adverse events"
Device defects checklist | through study completion, an average of one and a half year
  The risks to health and safety that may arise from the normal use of medical devices, including quality and malfunctions

CONTACTS AND LOCATIONS:
Overall Officials: Qinglong Gao, Principal Investigator — Zhejiang Fubon Technology Co., Ltd
Locations (1):
- Zhejiang Hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Xiong B, Wang X, Xu X, Lou Z, Tong T, Gu D, Zhang K, Liu H. Effectiveness and safety of a lower-limb walking assist device for motor function recovery in subacute stroke patients: A prospective, randomized, open, parallel-controlled, noninferiority study. J Int Med Res. 2025 Nov;53(11):3000605251396301. doi: 10.1177/03000605251396301. Epub 2025 Nov 20. PMID 41265879